CLINICAL TRIAL: NCT05113199
Title: Feasibility and Acceptability of Virtual Dignity Therapy for Palliative Care Patients With Advanced Cancer
Brief Title: Virtual Dignity Therapy for Palliative Care Patients With Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Deirdre R. Pachman, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-005065
Record Dates: First submitted 2021-08-30; First posted 2021-11-09 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Advanced Cancer
Keywords: Dignity Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual Dignity Therapy (Experimental)
  Interventions: Behavioral: Virtual Dignity Therapy

INTERVENTIONS:
Behavioral: Virtual Dignity Therapy — Virtual Dignity Therapy will be facilitated by a registered nurse or medical doctor trained in Dignity Therapy.

SUMMARY:
The purpose of this study is to determine if it is feasible and acceptable to recruit for and deliver the Virtual Dignity Therapy intervention to palliative care patients with advanced cancer.

DETAILED DESCRIPTION:
This study is an investigator-initiated, single site Mayo Clinic Rochester prospective minimal risk pilot study to determine feasibility and acceptability of Virtual Dignity Therapy. The Dignity Therapy intervention is a brief, individualized psychotherapy that aims to relieve psycho-emotional and existential distress and improve the experiences of patients whose lives are impacted by serious illness. This therapy offers patients an opportunity to reflect on their life with a trained facilitator and share their thoughts and memories with family and other people in their life. This therapy consists of a total of 3 sessions, with each session 2-4 weeks apart, in which the investigator provides questions focused on life review. The sessions are recorded and transcribed. The interventionist will work with patients to edit the document and provide a final generativity document for patient to keep and give to loved ones.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* English fluency
* No diagnosed dementia
* Diagnosis of advanced cancer
* Expected prognosis > 6 months
* Provide informed consent
* Ability to complete questionnaire(s) by themselves or with assistance

Exclusion Criteria:

* Other psychological co-morbidities such as untreated schizophrenia, bipolar disease
* Recent suicide attempt or psychiatric illness severe enough that hospitalization has been necessary in last 6 months
* Active delirium
* Participation in concurrent legacy offerings through the palliative care clinic

Inclusion Criteria for caregivers:

* Age ≥18 years
* English fluency
* Provide informed consent
* Supported patient through Dignity Therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Feasibility Number | 2 Years
  Study feasibility will be measured by the number of participants who enrolled and finished the study.
Acceptability | Week 8 (after 3rd intervention session)
  Acceptability, as measured by the 7-item Was it Worth It (WIWI Questionnaire).The questions are answered as either "yes, no, or uncertain," overall perception of quality of life change, overall perception of study experience, one open-ended feedback question, and an option to talk with someone about concerns. Positive responses indicate acceptability. Results are reported as individual items.

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Pachman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials